CLINICAL TRIAL: NCT02059655
Title: Prostaglandin F2-alpha Eye Drops (Bimatoprost) in Thyroid Eye Disease: a Randomised Controlled Double Blind Crossover Trial
Brief Title: Prostaglandin F2-alpha Eye Drops in Thyroid Eye Disease (Bima Study)
Acronym: BIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: National Institute for Social Care and Health Research (Unknown)
Responsible Party: Principal Investigator, Professor Colin Dayan, Professor, Cardiff University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPON 1266-14
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Graves' Ophthalmopathy
Keywords: Graves' disease
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease | interventions — Bimatoprost; Ophthalmic Solutions; Sodium Chloride; Potassium Chloride; borax; boric acid; Hydrochloric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye drop solution (Placebo Comparator): Patients will receive 1 dose daily over 3 month period followed by 2 months washout period. Subsequently patient will cross over to the opposite treatment and continue further treatment for 3 month period.
  Interventions: Drug: Eye drop solution
- Bimatoprost (Active Comparator): 1 drop daily of Bimatoprost 0.03%. Patients will receive 1 dose daily over 3 month period followed by 2 months washout period. Subsequently patient will cross over to the opposite treatment and continue further treatment for 3 month period.
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost
  Other Names: Trade Name Lumigan. MA number: EU/1/02/205/001-002. ATC Code: S01EE03
  Arms: Bimatoprost
Drug: Eye drop solution — Artificial tear drops
  Other Names: 1 drop daily; Hypromellose Ph Eur 0.3g in 100ml; Sodium chloride; Potassium chloride; Borax; Boric acid; Benzalkonium chloride solution; Purified water; Sodium hydroxide solution (to adjust pH); Hydrochloric acid
  Arms: Eye drop solution

SUMMARY:
The purpose of the study is to establish whether Bimatoprost eye drops are effective in reducing proptosis in inactive thyroid eye disease (TED) patients and improving quality of life in patients with TED. Current standard NHS treatment/care for inactive TED is artificial tears (used as the placebo in this study) or surgery if appropriate.

The IMP is Bimatoprost eye drops PGF2α (0.03%). This is already licensed eye drops usually used for glaucoma. Therefore the current trial's indication is outside its licenced indication. The Investigational Medicinal Product (IMP) will be used according to its licenced dosage and form. This is the first time that Bimatoprost will be used in the treatment of TED

DETAILED DESCRIPTION:
Thyroid eye disease (TED) is a chronic disfiguring and debilitating disease of the eyes which can lead to sight loss in severe cases. Patients with TED frequently have characteristic eyeball protrusion (proptosis) due to increased fat accumulation behind the eye. The discomfort and changes in appearance of the eyes is a source of severe psychological distress and impaired quality of life in many patients. Current treatments for TED are unsatisfactory and established non-surgical therapies which specifically reduce proptosis are lacking. Reduced eyelid protrusion has recently been reported as a side-effect of the use of prostaglandin analogue eye drops (e.g. Bimatoprost (PGF2-alpha)) in the routine treatment of glaucoma and we have laboratory data showing inhibition of fat cells by Bimatoprost. Hence PGF2-alpha eye drops potentially represent a simple, non-invasive low toxicity topical alternative to surgery in TED. However no clinical trials of Bimatoprost have been conducted in TED to date. The objective of this study is to determine whether Bimatoprost eye drops are effective in reducing proptosis and thus improving quality of life in patients with TED. Trial participants will be recruited from the TED clinic at the University Hospital Wales. The clinic is a regional referral centre for the treatment and study of TED and is run by a multidisciplinary team of ophthalmologists, endocrinologists, and orthoptists with expertise in TED. Following informed consent, participants will be randomised to receive Bimatoprost or placebo eye drops for three months after which they will undergo a two month drug washout period before switching to the opposite treatment in the final three months of study. The primary endpoint is a change in standardised measurements of proptosis while secondary endpoints will include changes in quality of life scores. This study will provide evidence for a novel application of bimatoprost in patients with TED.

ELIGIBILITY:
Inclusion Criteria:

1. Stable TED with no reported change in proptosis for at least 6 months. See section 4.1.1 for TED definition;
2. Clinical activity score <3 (Appendix 1);
3. Proptosis (subjective unilateral proptosis confirmed by asymmetry in exophthalmometry of >2mm OR greater than 20 mm on exophthalmometry measurement in one eye);
4. Euthyroid (thyroid function tests in the reference range);
5. If female, must be using a reliable form of contraception during the trial, e.g. oral contraceptive and condom, intra-uterine device (IUD) and condom, diaphragm with spermicide and condom.

Exclusion Criteria:

1. Age <18 yrs;
2. Dysthyroid optic neuropathy unless previously treated;
3. Pregnancy or lactation;
4. Previous Corneal Herpes Simplex infection;
5. On therapy for glaucoma or intraocular hypertension;
6. Less than 6 months from prior systemic steroid use;
7. Aphakia, pseudophakia with torn posterior lens capsule or anterior chamber lenses;
8. Patient with risk factors for cystoid macular oedema, iritis or uveitis;
9. Severe Asthma (risk of severe allergic reaction to medication);
10. Previous allergy to Bimatoprost or preservative.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be comparison of the change in ophthalmometry readings over the two 3 month treatment periods. | 1 year
  Reduction of 2 mm or more is regarded as clinically relevant

SECONDARY OUTCOMES:
Change in quality of life scores on the TED quality of life questionnaire (GO-QOL) | 1 year
  Whether there has been an improvement in patients' quality of life
Intraocular pressures | 1 year
  Whether there has been a change in intraocular pressures
Side effects | 1 year
  To consider the side effect profiles of Bimatoprost in TED patients during the study.
  Expected Adverse Reactions to the trial treatment(s) are detailed below:
  1. Commonly occurring cosmetic effects (approximate incidence)
     * Conjunctival redness (0.5%);
     * Lengthening of eyelashes - (average elongation 0.7mm);
     * Darkening of eye lashes (45-57%);
     * Peri-ocular skin pigmentation (3%);
     * Darkening of the iris (10.1%).
  2. Rare but potentially serious side effects (limited information available)
     * Iris cysts;
     * Cystoid macular oedema;
     * Anterior uveitis;
     * Reactivation of herpes simplex virus infection
Health economic outcomes | 1 year
  The primary intention of the economic evaluation is to explore the cost associated with TED treatment. In theory, Bimatoprost intervention would lead to the net cost savings to NHS in comparison to surgical rehabilitation that the patient otherwise will go through. We are aware of limitation in the trial design as this trial primary intention is to evaluate efficacy of Bimatoprost in TED, not to follow up patients until they might need surgery. However it would be useful to collect the resource use and quality of life data during this trial period on a pilot basis which may lead to a larger health economic focus study in the future. It is not envisaged that the crossover design will yield data that could allow a meaningful incremental cost-effectiveness ratio (ICER) to be calculated for Bimatoprost against placebo, as the duration of effects on perceived quality of life cannot be predicted in advance

CONTACTS AND LOCATIONS:
Overall Officials: Colin M Dayan, MA FRCP PhD, Principal Investigator — Cardiff University
Locations (1):
- University Hospital of Wales, Cardiff, Cardiff, United Kingdom